CLINICAL TRIAL: NCT06247722
Title: A Multinational, Prospective, Non-interventional Study, to Assess Real World Use of a Tocilizumab Biosimilar in Rheumatoid Arthritis Patients
Brief Title: Real World Use of Tocilizumab Biosimilar studY
Acronym: RUBY
Status: Active, not recruiting | Type: Observational
Sponsor: Fresenius Kabi SwissBioSim GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: TOCI-001-CNI
Record Dates: First submitted 2024-01-22; First posted 2024-02-08 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Rheumatoid Arthritis
Keywords: tocilizumab; rheumatoid arthritis; persistence; real world use; biosimilar; biosimilar switch; Tyenne
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this non interventional study is to evaluate the use of Tyenne, a tocilizumab biosimilar, in a real world setting in Rheumatoid Arthritis (RA) patients over a period of 12 months.

The main questions it aims to answer are:

* What is the patients' persistence on Tyenne (patient's ability to continue the treatment for the prescribed duration), 6 months after treatment start?
* What is the patients' persistence on Tyenne (patient's ability to continue the treatment for the prescribed duration), 12 months after treatment start?

The decision of prescribing Tyenne will be done by the physician independently, prior to patient enrolment in the study. Enrolled patients will be followed for 12 months following Tyenne treatment start, or until they permanently discontinue Tyenne.

There will be one baseline visit and three follow-up visits at approximately 3, 6 and 12 months after Tyenne treatment initiation. All follow-up visits will be conducted according to the physician current clinical practice and are not imposed due to this protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients initially diagnosed with moderate to severe rheumatoid arthritis (RA) according to ACR/EULAR 2010 rheumatoid arthritis classification criteria
* Patients for whom the decision to prescribe Tyenne, a tocilizumab biosimilar has been made by the investigator prior to the inclusion, in accordance with the Summary of Product Characteristics (SmPC), local label and physician' current clinical practice
* Patients able to understand and complete the study questionnaires in local language during the study visits
* Patients are willing to enter the study (signed informed consent)

Exclusion Criteria:

* Patients participating or expected to participate in any interventional clinical trial during their treatment with Tyenne, a tocilizumab biosimilar

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include male and female adult patients with moderate to severe rheumatoid arthritis (RA) who
  * were prescribed Tyenne, a tocilizumab biosimilar
  * meet all the study inclusion criteria
  * meet none of the exclusion criteria
  * provide written informed consent to participate.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2026-03-05 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Persistence of tocilizumab treatment 6 months after treatment start with Tyenne, a tocilizumab biosimilar | 6 months after treatment start
  A patient is considered to still be on tocilizumab biosimilar treatment (persistence equal "Yes") if no permanent discontinuation of the tocilizumab biosimilar treatment and no lost to follow-up is reported by the investigator before the visit. A patient will be considered to have discontinued the tocilizumab biosimilar (not persistent) at 6 month timepoint if a) the investigator reports a permanent discontinuation of the treatment before the timepoint or b) the patient is lost to follow-up at the timepoint. Temporary cessations of the biosimilar will not be considered as treatment discontinuation, and the treatment will be considered persistent.

SECONDARY OUTCOMES:
Persistence of tocilizumab treatment 12 months after treatment start with Tyenne, a tocilizumab biosimilar | 12 months after treatment start
  A patient is considered to still be on tocilizumab biosimilar treatment (persistence equal "Yes") if no permanent discontinuation of the tocilizumab biosimilar treatment and no lost to follow-up is reported by the investigator before the visit. A patient will be considered to have discontinued the tocilizumab biosimilar (not persistent) at 12 month timepoint if a) the investigator reports a permanent discontinuation of the treatment before the timepoint or b) the patient is lost to follow-up at the timepoint. Temporary cessations of the biosimilar will not be considered as treatment discontinuation, and the treatment will be considered persistent.
Change from Baseline in Disease Activity Score 28 (DAS28-ESR or DAS 28-CRP) at Month 12 | 12 months after treatment start
Change from Baseline in Patient Global Assessment of Disease Activity at Month 12 | 12 months after treatment start
Change from Baseline in Physician Global Assessment of Disease Activity at Month 12 | 12 months after treatment start

CONTACTS AND LOCATIONS:
Locations (8):
- Germany (8):
  - Rheumatologische Schwerpunktpraxis Berlin, Berlin
  - Rheumapraxis Dr. Liebhaber Halle, Halle
  - Facharztpraxis für Innere Medizin Ludwigsfelde, Ludwigsfelde
  - Rheumatologische Facharztpraxis, Magdeburg
  - Facharztpraxis für Innere Medizin, Naumburg
  - Klinische Forschung, Planegg
  - Rheumahaus Potsdam, Potsdam
  - Rheumatologische Facharztpraxis Templin, Templin

IPD SHARING:
Plan to Share IPD: No